CLINICAL TRIAL: NCT04683250
Title: Phase I/II Study of the Selective RET Inhibitor TAS0953/HM06 in Patients with Advanced Solid Tumors with RET Gene Abnormalities
Brief Title: Study of RET Inhibitor TAS0953/HM06 in Patients with Advanced Solid Tumors with RET Gene Abnormalities
Acronym: MARGARET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM06-19-26
Record Dates: First submitted 2020-12-04; First posted 2020-12-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: RET-altered Non Small Cell Lung Cancer; RET-altered Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose escalation phase followed by a dose expansion phase (Phase 1), then followed by a Phase 2 at the recommended dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAS0953/HM06 Phase 1 (Experimental): Dose escalation and dose expansion until recommended Phase 2 dose determined
  Interventions: Drug: TAS0953/HM06
- TAS0953/HM06 Phase 2 (Experimental): Treatment phase at recommended Phase 2 dose in three different populations
  Interventions: Drug: TAS0953/HM06

INTERVENTIONS:
Drug: TAS0953/HM06 — Phase 1: oral, starting dose 20mg twice a day, until recommended phase 2 dose, continuous daily dosing, cycles lasting 21 days
  Arms: TAS0953/HM06 Phase 1
Drug: TAS0953/HM06 — Phase 2: oral, recommended dose twice a day, continuous daily dosing, cycles lasting 21 days
  Arms: TAS0953/HM06 Phase 2

SUMMARY:
Phase 1 and 2 trial to study the safety, pharmacokinetics, and efficacy of TAS0953/HM06 in patients with advanced solid tumors with RET gene abnormalities. Phase 1 aims to determine the Maximum Tolerated Dose (MTD) and identify the Recommended Phase 2 Dose (RP2D) to be used in phase 2.

ELIGIBILITY:
Inclusion Criteria:

Phase I - Common inclusion criteria for Dose-Escalation / Dose-Expansion:

* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Available RET-gene abnormalities determined on tissue biopsy or liquid biopsy. If deemed appropriate by the investigator, determination on a pleural cell block is also acceptable.
* Adequate hematopoietic, hepatic and renal function

Phase I Dose-Escalation - Specific inclusion criteria:

* Advanced solid tumors
* Measurable and/or non-measurable disease as determined by RECIST 1.1
* If patient has brain and/or leptomeningeal metastases, (s)he should be asymptomatic.

Phase I Dose-Expansion - Specific inclusion criteria:

* Patient with RET gene fusion :

  * Cohort 1, 3: locally advanced or metastatic NSCLC patients naïve to RET selective inhibitors and no prior systemic anti-cancer treatment. Patients who have been treated with neo-adjuvant or adjuvant chemotherapy may be included if it has been completed at least 6 months prior to the first dose of the study.
  * Cohort 2, 4: locally advanced or metastatic NSCLC patients with RET gene fusion and prior exposure to RET selective inhibitors.
* Measurable disease as determined by RECIST 1.1
* If patient has brain and/or leptomeningeal metastases,(s)he should have:

  * asymptomatic untreated brain/leptomeningeal metastases off steroids and anticonvulsant for at least 7 days or
  * asymptomatic brain metastases already treated with local therapy and be clinically stable on steroids and anticonvulsant for at least 7 days before study drug administration.

Phase II :

* Available RET-gene abnormalities determined on tissue or liquid biopsy
* Locally advanced or metastatic:

  * NSCLC patients with primary RET gene fusion and prior exposure to RET selective inhibitors;
  * NSCLC patients with RET gene fusion and without prior exposure to RET selective inhibitors
  * patients with advanced solid tumors that harbour RET gene abnormalities (other than NSCLC patients with primary RET gene fusions) and has failed all the available therapeutic options
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Measurable disease as determined by RECIST 1.1
* If patient has brain and/or leptomeningeal metastases,(s)he should have:

  * asymptomatic untreated brain/leptomeningeal metastases off steroids and anticonvulsant for at least 7 days or
  * asymptomatic brain metastases already treated with local therapy and be clinically stable on steroids and anticonvulsant for at least 7 days before study drug administration.
* Adequate hematopoietic, hepatic and renal function

Exclusion Criteria:

Common exclusion criteria for Phase 1 and Phase 2

* Investigational agents or anticancer therapy within 5 half-lives prior to the first dose of study drug
* Major surgery (excluding placement of vascular access) within 4 weeks prior to the first dose of study drug or planned major surgery during the course of study treatment.
* Whole Brain Radiotherapy within 14 days or other palliative radiotherapy within 7 days prior to the first dose of study drug, or persisting side effects of such therapy, in the opinion of the Investigator.
* Clinically significant, uncontrolled, cardiovascular disease including myocardial infarction within 3 months prior to Day 1 of Cycle 1, unstable angina pectoris, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic Congestive Heart Failure (CHF) New York Heart Association (NYHA) class III-IV, and severe uncontrolled arterial hypertension, according to the Investigator's opinion.
* QT interval corrected using Fridericia's formula (QTcF) >470 msec; personal or family history of prolonged QT syndrome or history of Torsades de pointes (TdP). History of risk factors for TdP
* Treatment with strong CYP3A4 inhibitors within 1 week prior to the first dose of study drug or strong CYP3A4 inducers within 3 weeks prior to the first dose of study drug.

Phase I Dose-Expansion - and Phase II specific exclusion criteria:

* Presence of known EGFR, KRAS, ALK, HER2, ROS1, BRAF and METex14 activating mutations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (dose-escalation): Maximum Tolerated Dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  Incidence rate and category of dose limiting toxicities (DLTs)
Phase 1 (dose-expansion): Recommended Phase 2 dose (RP2D) | At the end of Cycle 1 (each cycle is 21 days), and at the end of every subsequent cycle (each cycle is 21 days) for approximately 10 months (or earlier if patient discontinues the study)
Phase 2: Objective Response Rate (ORR) by independent central review | Approximately every 6 weeks for 6 months, then every 9 weeks during treatment, 7 days after the last dose, and every 3 months after the last dose (up to an average of 2 years) in patients without progressive disease.
  Proportion of patients with confirmed complete response (CR) and or partial response (PR) according to RECIST 1.1 as assessed by independent central review

SECONDARY OUTCOMES:
Phase 1 (dose expansion): Objective Response Rate (ORR) by independent central review | Approximately every 6 weeks for 6 months, then every 9 weeks during treatment, 7 days after the last dose, and every 3 months after the last dose (up to an average of 2 years) in patients without progressive disease
  Proportion of patients with confirmed complete response (CR) and or partial response (PR) according to RECIST 1.1 as assessed by independent central review
Phase 2: ORR by Investigator | Approximately every 6 weeks for 6 months, then every 9 weeks during treatment, 7 days after the last dose, and every 3 months after the last dose (up to an average of 2 years) in patients without progressive disease
  Proportion of patients with confirmed complete response (CR) and or partial response (PR) according to RECIST 1.1 as assessed by Investigator
Phase 2: Disease Control Rate (DCR) | Approximately every 6 weeks for 6 months, then every 9 weeks during treatment, 7 days after the last dose, and every 3 months after the last dose (up to an average of 2 years) in patients without progressive disease
  Proportion of patients with confirmed complete response (CR), partial response (PR) and Stable Disease according to RECIST 1.1 as assessed by Investigator
Phase 2: Time to Tumor Response (TTR) | From date of randomization until the date of first documentation of objective tumor response, assessed up to an average of 2 years.
  Time from first dose to first documentation of objective tumor response (CR or PR)
Phase 2: Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or death due to any cause, whichever occurs first, assessed up to an average of 2 years.
  Time from first dose to first documentation of objective disease progression or to death due to any cause, whichever occurs first
Phase 2: Time to Progression (TTP) | From date of randomization until the date of first documented progression, assessed up to an average of 2 years
  Time from first dose to objective tumor progression
Phase 2: Duration of Response (DOR) | From first documentation of objective tumor response (CR or PR) until the date of first documented progression or death due to any causes, whichever occurs first, assessed up to an average of 2 years
  Time from first documentation of tumor response (CR + PR) to disease progression or death due any cause whichever occurs first
Phase 2: Overall Survival (OS) | From date of randomization until the date of death due to any cause, assessed up to an average of 2 years
  Time from first dose to date of death due to any cause
Phase 2: Central Nervous System (CNS) ORR (C-ORR) | Approximately every 6 weeks for 6 months, then every 9 weeks during treatment, 7 days after the last dose, and every 3 months after the last dose (up to an average of 2 years) in patients without progressive disease
  Rate of confirmed CR and PR relative to patients with brain lesions at study entry
Phase 2: Central Nervous System DOR (C-DOR) | From first documentation of objective tumor response (CR or PR) until the date of first documented progression or death due to any causes, whichever occurs first, assessed up to an average of 2 years
  Time from documentation of intracranial tumor response to disease progression or death due to any cause whichever occurs first
Phase 2: Time to CNS progression | From date of randomization until the date of first documented progression, assessed up to an average of 2 years
  Time from the first dose to the first radiological evidence of CNS disease progression
Phase 1 (dose-escalation): Area under the plasma concentration versus time curve from time 0 to 12 hours (AUC0-12) | Day -1 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): AUC0-24 | Day -1 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): AUC0-infinity | Day -1 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): AUC0-12 at steady state | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Maximum drug concentration (Cmax) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Trough drug concentration at 12 hours (Ctrough) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Time to maximum plasma concentration (tmax) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Terminal half-life (t1/2) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Accumulation factor based on Cmax (Rmax) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Accumulation factor based on Ctrough (Rmin) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Terminal rate constant (lambda_z) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Volume of Distribution (Vz/F) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Systemic clearance (CL/F) | Day -1 and Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Amount excreted in 0-24 hour urine (Ae0-24) | Day -1 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-escalation): Renal Clearance (CL_R) | Day -1 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): AUC0-12 at steady state | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): Maximum drug concentration (Cmax) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): Trough drug concentration at 12 hours (Ctrough) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): Time to maximum plasma concentration (tmax) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): Terminal rate constant (lambda_z) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1 (dose-expansion): Terminal half-life (t1/2) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 2 Population PK: Typical value of absorption rate constant (Ka) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 2 Population PK: Typical value of CL/F | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 2 Population PK: Typical value of volume of distribution (V/F) | Day 15 of Cycle 1 (each cycle is 21 days)
Phase 1: Incidence of abnormal electrocardiograms (ECG QT interval). QT will be corrected for heart rate (QTc) using Fridericia's formula (QTcF). | On Day 1, Day 8 (only in dose escalation), Day 15 in cycle 1, Day 1 of any subsequent cycles (each cycle is 21 days) during treatment, for approximately 10 months (or earlier if the patient discontinues from the study), and 7 days after last dose
Phase 1: Incidence of treatment-emergent adverse events (TEAEs) | From the time of informed consent, for approximately 10 months (or earlier if the patient discontinues from the study), and through Safety Follow-up (28 days after the last dose)
Phase 1: Incidence of serious adverse events (SAEs) | From the time of informed consent, for approximately 10 months (or earlier if the patient discontinues from the study), and through Safety Follow-up (28 days after the last dose)
Phase 2: Incidence of abnormal electrocardiograms (ECG QT interval). QT will be corrected for heart rate (QTc) using Fridericia's formula (QTcF). | On Day 1 and Day 15 in cycle 1, Day 1 of any subsequent cycles (each cycle is 21 days) during treatment, for approximately 2 years (or earlier if the patient discontinues from the study), and 7 days after last dose
Phase 2: Incidence of treatment-emergent adverse events (TEAEs) | From the time of informed consent for approximately 2 years (or earlier if the patient discontinues from the study), and through Safety Follow-up (28 days after the last dose)
Phase 2: Incidence of serious adverse events (SAEs) | From the time of informed consent for approximately 2 years (or earlier if the patient discontinues from the study), and through Safety Follow-up (28 days after the last dose)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - START Midwest - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
- Japan (8):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Shunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided